CLINICAL TRIAL: NCT05557812
Title: A Comparative Assessment Clinical Trial Comparing Ferric Sulfate With Zinc-oxide Eugenol and Non-eugenol Based Materials for Pulpotomy in Primary Molar Teeth
Brief Title: A Clinical Trial Comparing FS With ZOE and Non-eugenol Based Materials in Primary Teeth Pulpotomies
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20024506
Record Dates: First submitted 2022-09-07; First posted 2022-09-28 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Pulpitis
MeSH Terms: conditions — Pulpitis | interventions — ferric sulfate; Cavit

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- non-eugenol based ZOE and Ferric Sulfate (Experimental): non-eugenol based ZOE and Ferric Sulfate in primary molar pulpotomy procedures.
  Interventions: Drug: non-eugenol based ZOE base material with Ferric Sulfate in primary molar pulpotomies
- eugenol based zinc oxide and Ferric Sulfate (Experimental): eugenol based zinc oxide and Ferric Sulfate in primary molars pulpotomies procedures.
  Interventions: Drug: eugenol based zinc oxide and Ferric Sulfate

INTERVENTIONS:
Drug: non-eugenol based ZOE base material with Ferric Sulfate in primary molar pulpotomies — non-eugenol based ZOE base material placed over ferric sulphate, during vital pulp therapy (pulpotomy) in primary molars
  Other Names: CAVIT
  Arms: non-eugenol based ZOE and Ferric Sulfate
Drug: eugenol based zinc oxide and Ferric Sulfate — eugenol based zinc oxide base material placed over Ferric Sulfate medicament, during vital pulp therapy (pulpotomy) in primary molars
  Other Names: Intermediate Restorative Material (IRM)
  Arms: eugenol based zinc oxide and Ferric Sulfate

SUMMARY:
Internal resorption in the most common cause of failure in FS pulpotomies in primary molars. This has been attributed to the release of free eugenol from the zinc and eugenol mixture of the base material over the pulp tissue. Zinc oxide-eugenol (ZOE) paste is the most common base material placed over the infected pulp tissues during pulpotomies of primary molars, however the evidence suggests that the eugenol component has been associated with the failure of the vital pulp treatment in primary molars. Cavit (3M, US) is another base material that contains Zinc-oxide, zinc sulphate, and calcium salts without eugenol. The effectiveness of non-eugenol based Zinc oxide as a base material over ferric sulphate treated pulp has not been explored. The hypothesis is that the non-eugenol based ZOE could be used as an alternate to eugenol based ZOE and thereby avoid the radiological failures. Therefore, this randomized controlled clinical split-mouth trial aimed to evaluate and compare the effect of eugenol and non-eugenol based ZOE on the success of primary tooth pulpotomies where FS is used as a medicament.

DETAILED DESCRIPTION:
Pulpotomy vital pulp therapy is a frequently performed therapeutic procedures in pediatric dentistry. This procedure aims to preserve the vitality of primary teeth or immature permanent teeth with pulp exposure due to caries and with no evidence of radiographical pathology. Pulpotomies eliminate the bacterial infection from the tooth by the partial removal of the apical pulp tissue, followed by the placement of a pulp medicament and a base material on top of it. The most frequently used medicaments in pulpotomy vital therapy are formocresol (FC), mineral trioxide aggregate (MTA), ferric sulphate (FS), calcium hydroxide (CH), Bio-dentine (BD) and laser. Due to its high success rate, FC is a commonly used medicament, and it is described as the 'gold standard' for pulpotomy procedures. However, FC is a controversial medicament, because ethe major component of formocresol; formaldehyde, has been classified by the International Agency for Research on Cancer (IARC) as a possible human carcinogen. Consequently, several studies were conducted to assess the toxic effects of using FC, and the evidence suggested that, in the dental setting, there is very low exposure of formaldehyde, and it should not exhibit any carcinogenic actions. Despite these findings dentists in Europe still have some concerns regarding FC usage in vital pulp therapy, and alternatively prefer other medicaments over FC, Such as Ferric Sulfate (FS); which is their medicament of choice. FS is a hemostatic agent that is commonly used for pulpotomies in primary teeth, this agent helps in retaining the vitality of the tooth by forming a protective metal protein clot over the vital pulp tissue. Therefore, FS has been widely studied over the world, and the evidence suggested that both FC and FS showed comparable success rates clinically and radiographically as medicaments for pulpotomies in primary molars. However, FC was anticipated to achieve a 10% higher success over FS in a Trial Sequential Analysis (TSA) that was conducted at 24 months' time interval comparing the radiographic success of FC and FS. These finding can be explained by the fact that internal resorption in the most common cause of failure in FS pulpotomies in primary molars. This has been attributed to the release of free eugenol from the zinc and eugenol mixture of the base material over the pulp tissue. Zinc oxide-eugenol (ZOE) paste is the most common base material placed over the infected pulp tissues during pulpotomies of primary molars, however the evidence suggests that the eugenol component has been associated with the failure of the vital pulp treatment in primary molars. Cavit (3M, US) is another base material that contains Zinc-oxide, zinc sulphate, and calcium salts without eugenol. This has been used a temporary restorative material with excellent sealing capability. It has been shown that this material induces an alkaline potential hydrogen (pH), which in terms plays an important role in hard tissue formation, by the neutralization of the lactic acid formation from osteoclasts and the activation of the alkaline phosphatases. The effectiveness of non-eugenol based Zinc oxide as a base material over ferric sulphate treated pulp has not been explored. The hypothesis is that the non-eugenol based ZOE could be used as an alternate to eugenol based ZOE and thereby avoid the radiological failures. Therefore, this randomized controlled clinical split-mouth trial aimed to evaluate and compare the effect of eugenol and non-eugenol based ZOE on the success of primary tooth pulpotomies where FS is used as a medicament.

Null hypothesis: In primary molar pulpotomy, non-eugenol based ZOE placed over ferric sulphate do not show higher success rate compared to eugenol based zinc oxide as a base material

Alternate hypothesis: In primary molar pulpotomy, non-eugenol based ZOE placed over ferric sulphate show a higher success rate compared to eugenol based zinc oxide as a base material

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 7 years old.
* Carious teeth with clinical and radiographic diagnosis of reversible pulpitis
* Only teeth having no more than one third of their roots undergoing physiologic resorption were included.
* Restorable with stainless steel crown

Exclusion Criteria:

* clinical or radiographic evidence of pulp degeneration
* excessive bleeding
* pathologic mobility
* swelling or fistula
* history of spontaneous and nocturnal pain
* tenderness to percussion or palpation
* external or internal root resorption : {The primary teeth undergo resorption due to developing permanent teeth which is considered normal. Presence of internal root resorption will be considered as a failure (pathological change). Alternatively external root resorption will not be considered as a failure (physiological change}
* inter radicular or periapical radiolucency.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Clinical success rate | 36 months
  The pulpotomy procedure was considered clinically successful if there were no pain, swelling, tenderness to percussion, abscess or abnormal mobility.
Radiographic success rate | 36 months
  1. Normal periodontal ligament space
  2. No inter-radicular or periapical radiolucency
  3. No internal or external root resorption

CONTACTS AND LOCATIONS:
Overall Officials: Jayakumar Jayaraman, BDS MDS PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No